CLINICAL TRIAL: NCT04287348
Title: Intravitreal Brolucizumab in Neovascular Age-related Macular Degeneration With Limited Response to Aflibercept
Acronym: ROBIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to safety letter beovu from Novartis
Sponsor: Vista Klinik (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, PD Dr. med. Katja Hatz, Head of Medical Retina and clinical Research department, Vista Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROBIN / CRTH258ACH01T
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD, poor responders, aflibercept, brolucizumab
MeSH Terms: interventions — brolucizumab; Solutions; Intravitreal Injections

STUDY DESIGN:
Intervention Model Description: Prospective, one-treatment-arm, monocentre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Beovu (Brolucizumab) (Other): Prospective, one-treatment-arm, monocentre study
  Interventions: Drug: Brolucizumab 6 mg solution for intravitreal injection

INTERVENTIONS:
Drug: Brolucizumab 6 mg solution for intravitreal injection — All consenting, enrolled patients (irrespectively of maximum recurrence-free interval under aflibercept pretreatment) will receive an intravitreal injection of brolucizumab 6 mg at baseline (week 0), at week 4 and each of the following treat and extend visits. At each visit all patients will undergo an OCT assessment. For all patients extension of treatment intervals is only possible 2-week-stepwise, e.g. 4, 6, 8 weeks etc.
  Other Names: Beovu

SUMMARY:
The purpose of this investigator initiated study is to identify the effects of intravitreal brolucizumab on recurrence-free treatment intervals and morphological features in choroidal neovascularizations (CNV) due to age-related macular degeneration (AMD) in which the Optical coherence tomography (OCT) guided treatment interval failed to be extended to 6, 8 or 10 weeks intervals in a treat and extend regimen using aflibercept.

DETAILED DESCRIPTION:
Outcome Measures:

The primary outcome is the mean maximum treatment interval with intravitreal brolucizumab at month 6 and 12.

The secondary outcomes are:

* Best corrected visual acuity (BCVA) in letters and BCVA change (letters) from baseline (=switch to brolucizumab) to month 6 and 12.
* Number of brolucizumab intravitreal treatments applied during the 12 months study period.
* Central retinal thickness (CRT, in µm) as measured in the central ETDRS subfield Spectral-Domain Optical coherence tomography (SD-OCT) at baseline, month 6 and 12.
* Presence of qualitative SD-OCT features like intraretinal fluid, subretinal fluid, pigment epithelial detachment and hyperreflective foci at baseline, month 6 and 12.
* Total CNV area and vessel density as measured by OCTangiography (OCTA) at baseline, month 6 and 12.
* Total area of leakage from CNV and the total lesion area as evaluated by Fluorescein angiography (FA) at baseline and month 12.
* VFQ-25 total and subscores as evaluated by quality of life questionnaire VFQ-25 at baseline and month 6 and 12.
* Rates of adverse events and serious adverse events at 6 and 12 months.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥ 50 years of age.
* Patients with active subfoveal or juxtafoveal Type 1, 2 or 3 CNV secondary to AMD.
* Pre-treatment with intravitreal aflibercept in a treat and extend regimen with 2-weeks steps and failing to be extended by two weeks to either 6-weeks intervals, 8 week intervals or 10 week intervals without showing CNV activity (at least 2 attempts to extend).
* The total area of CNV (including both classic and occult components) encompassed within the lesion must be ≥ 50% of the total lesion area.
* The total lesion area ≤ 12 disc areas for minimally classic or occult with no classic component and ≤ 9 disc areas (5400μm) in greatest linear dimension with predominantly classic lesions.
* Patients who have a BCVA of at least 20/160 (letter score 40 letters) in the study eye using ETDRS charts.
* Willing and able to give written informed consent according to legal requirements, and who have signed the consent form prior to initiation of any study procedure including withdrawal from exclusionary medications for the purpose of this study.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either ≥ 50% of the total lesion area or ≥ 1 disc area in size.
* Presence of a retinal pigment epithelial tear involving the fovea in the study eye.
* Patients with angioid streaks or precursors of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia.
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the 12 months study period.
* Vitreous hemorrhage or history of retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Active intraocular inflammation (grade trace or above) in the study eye.
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as idiopathic or autoimmune-associated uveitis in either eye.
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication).
* Aphakia with absence of the posterior capsule in the study eye.
* Any prior treatment in the study eye with radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, transpupillary thermotherapy.
* History of submacular surgery or other surgical intervention for AMD in the study eye, glaucoma filtration surgery, corneal transplant surgery.
* Extracapsular extraction of cataract with phacoemulsification within three months preceding Baseline, or a history of post-operative complications within the last 12 months preceding Baseline in the study eye (uveitis, cyclitis, etc.).
* Use of other investigational drugs at the time of baseline, or within 30 days or 5 half- lives of baseline, whichever is longer (excluding vitamins and minerals).
* Previous violation of the posterior capsule in the study eye unless it occurred as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml).
* History of hypersensitivity or allergy to fluorescein.
* Inability to obtain OCTs, OCTAs, fundus photographs or fluorescein angiograms of sufficient quality.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the mean maximum treatment interval with intravitreal brolucizumab at month 6 and 12. | up to month 12
  mean maximum treatment interval with intravitreal brolucizumab

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) in letters | month 6 and 12
  BCVA
Number of brolucizumab intravitreal treatments applied during the 12 months study period. | 12 months
  Number of brolucizumab
Central retinal thickness (CRT, in µm) as measured in the central ETDRS subfield Spectral-Domain Optical coherence tomography (SD-OCT) at baseline, month 6 and 12. | month 6 and 12
  CRT
Presence of qualitative SD-OCT features like intraretinal fluid, subretinal fluid, pigment epithelial detachment and hyperreflective foci at baseline, month 6 and 12 | month 6 and 12
  SD-OCT
Total CNV area and vessel density as measured by OCTangiography (OCTA) at baseline, month 6 and 12. | month 6 and 12
  Total CNV area and vessel density
Total area of leakage from CNV | baseline and month 12
  Total area of leakage from CNV
VFQ-25 total evaluated by quality of life questionnaire VFQ-25 at baseline and month 6 and 12. | month 6 and 12
  VFQ-25
Rates of adverse events and serious adverse events at 6 and 12 months. | 6 and 12 months.
  AE and SAE
BCVA change (letters) from baseline (=switch to brolucizumab) | month 6 and 12
  BCVA
the total lesion area as evaluated by Fluorescein angiography (FA) at baseline and month 12 | baseline and month 12
  Total area of leakage from CNV
VFQ-25 subscores | month 6 and 12
  VFQ-25 subscores

CONTACTS AND LOCATIONS:
Overall Officials: Katja Hatz, PD Dr. med, Principal Investigator — Vista Klinik Binningen
Locations (1):
- Vista Klinik, Binningen, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No